CLINICAL TRIAL: NCT03010371
Title: Presential Vs Online Group-based Psychosocial Treatment for Breast Cancer Survivors: A Multicentre Randomised Controlled Trial. Efficacy, Medical Cost Offset and Treatment Predictors.
Brief Title: Presential Vs Online Group-based Psychosocial Treatment for Breast Cancer Survivors.
Acronym: PSONLINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Català d'Oncologia (Other)
Responsible Party: Principal Investigator, Cristian Ochoa Arnedo, PhD, Institut Català d'Oncologia
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ICOLH201601
Record Dates: First submitted 2016-12-18; First posted 2017-01-05 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Breastcancer; Emotional Disorder; Distress
Keywords: positive psychotherapy, online, breast cancer, survivors
MeSH Terms: conditions — Breast Neoplasms | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The current clinical trial is a sequential RCT. In the first stage, it compares the effectiveness of the Positive Psychotherapy for Cancer with one of the most proved Cognitive-Behavioral Psychotherapies in Cancer, which is the Cognitive Behavioral Stress Management (CBSM). In the other stage, the common presential version of the Positive Psychotherapy is compared with its online version.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Positive Psychotherapy (Experimental): A group of breast cancer survivors are randomly allocated to the presential version of the positive psychotherapy
  Interventions: Behavioral: Positive Psychotherapy
- Positive Online Psychotherapy (Experimental): A group of breast cancer survivors are randomly allocated to the online version of the positive psychotherapy
  Interventions: Behavioral: Positive Online Psychotherapy
- Cognitive Behavioral Therapy (Experimental): A group of breast cancer survivors are randomly allocated to the presential cognitive behavioral therapy (Cognitive Behavioral Stress Management, CBSM)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Positive Psychotherapy — Positive Psychotherapy (PP) is designed to treat cancer survivors with moderate/severe adaptation difficulties after completing cancer treatments (Ochoa et al., 2010). The objectives are the facilitation and promotion of post-traumatic growth and quality of life, and the reduction of emotional distress (anxiety, depression and post-traumatic symptoms). Secondary consequences of this psychological improvement is a better transition to daily life and the restoration of a good psychosocial functioning (labor reincorporation, adherence to treatments and follow-up, and the adoption of healthy lifestyles). The program consists of twelve sessions of 90 minutes per week in a closed group (5 to 7 participants). Each session focuses on the different topics and tasks defined in the Positive Psychotherapy for cancer survivors (Ochoa et al., 2010).
  Arms: Positive Psychotherapy
Behavioral: Positive Online Psychotherapy — The Positive Online Psychotherapy (POP) is based on the PP program, but being adapted to an online version. Patients in this experimental condition will have access to a secure virtual platform (supervised and dependent from the Catalan Health Department). The POP consists of twelve weekly sessions of 90 minutes, in a closed-group format (5-7 participants). Patients have a simultaneous group-connection to the online platform, together with a clinical psychologist who lead the tasks according to the focuses of each session.
  Arms: Positive Online Psychotherapy
Behavioral: Cognitive Behavioral Therapy — The Cognitive Behavioral Therapy (CBT) is based on the Cognitive Behavioral Stress Management (Antoni, 2003) and the training program derived from it, "Breast Cancer Stress Management and Relaxation Training" (B-SMART) by Antoni Michael (2003). In its Spanish version, it is a 10-session therapy aimed to reduce cancer-related emotional distress, facilitating adjustment to illness and greater quality of life. Stress management and relaxation techniques help patients to identify their own stress responses and learn alternative ways of thinking and acting in response to the demands they perceive as highly stressful.
  Arms: Cognitive Behavioral Therapy

SUMMARY:
This multicenter study is a sequential RCT which aims to prove, in the first stage, the efficacy of a face-to-face Positive Psychotherapy in Cancer (PPC) group compared to a Cognitive Behavioral Stress Management (CBSM) group. In the second stage, the common face-to-face version of the PPC will be compared with its online version via videoconference (Online group Positive Psychotherapy, OPPC) among a group of primary breast cancer survivors. The principal dependent variables assessed will be emotional distress, post-traumatic growth (PTG) and quality of life (QoL). Some treatment predictors of psychosocial response will be explored. Lastly, an economic analysis focused on the Quality Adjusted Life Years (QALY) will be carried out at each stage. For the first stage, we hypothesize that the PCC group would achieve similar efficacy in reducing participants' distress compared to the CBSM group, while the PCC group would show greater improvement in PTG than the CBSM group. For the second stage, it is hypothesized that the OPCC would achieve similar efficacy in all psychosocial variables and guarantee equivalent retention and adherence compared to face-to-face PPC.

DETAILED DESCRIPTION:
Psychosocial treatments in cancer survivors have demonstrated their efficacy in reducing emotional distress and improving Quality of Life (QoL). Providing access to a psychosocial intervention at the end of a curative cancer treatment becomes worthwhile, not only because it reduces the use of other medical resources and promotes return-to-work, but also because it facilitates oncological treatment adherence and the adoption of healthy lifestyles. Online psychosocial treatments are a good option because of their easy access, anonymity and low cost. The study is a sequential multicenter, controlled and randomized clinical trial organized in two stages. It is worth highlighting that there was a deviance from the initial research plan which contemplated a three-arm clinical trial. However, during the preparation of the recruitment phase, we faced some problems related to the opening of the third arm (online group positive psychotherapy) due to the fact that the required technology that supported the online group psychotherapy was not available for use at that moment. As a result, we decided to wait for a few months before we activate the third arm of the study. In conclusion, the study aims to prove, in the first stage, the efficacy of a face-to-face Positive Psychotherapy in Cancer (PPC) group compared to a Cognitive Behavioral Stress Management (CBSM) group. In the second stage, the common face-to-face version of the PPC will be compared with its online version via videoconference (Online group Positive Psychotherapy, OPPC). Those breast cancer survivors who have showed moderate or severe adaptation problems after the completion of their oncological treatment will be randomly assigned to PPC versus CBSM group for the first stage of the study (January 2013-December 2015), and for the second stage, a different group of breast cancer survivors will be assigned to PPC versus OPCC (January 2016-February 2019). Regarding the methodology of the study, participants from the 4 groups will be evaluated using a battery of measures at the beginning of the study (T0), post-treatment (T1), 3 months from T1 (T2) and 12 months from T2 (T3). Therefore, this study will use a factorial design of 3 (treatment conditions) x 4 (evaluation points).The main outcome measures include: quality of life, anxiety, depression, post-traumatic stress and post-traumatic growth. Secondary outcome measures will be: healthy lifestyles, adherence to the oncological treatment, perceived social support, and the number of return-to-work days after the cancer treatment completion.

Data will be analyzed using SPSS 21.0 version. For the first stage, we hypothesize that the PCC group would achieve similar efficacy in reducing participants' distress compared to the CBSM group, while the PCC group would show greater improvement in PTG. For the second stage, it is hypothesized that the OPCC would achieve similar efficacy in all psychosocial variables and guarantee equivalent retention and adherence compared to face-to-face PPC. Besides, the presential format will be more effective for severely distressed patients with previous history of trauma, while the online format will be more effective for younger patients with mild emotional distress.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary breast cancer,
* Having completed the curative treatment and / or adjuvant treatment for their primary tumor in the last 1 to 6 months
* Be able to use the Internet in a private place and have a knowledge of Internet at the user level
* Scoring ≥ 5 points on the thermometer for emotional distress (anxiety and depression) and confirmed with a score on the HADS total scale ≥ 10 in the admission interview.

Exclusion Criteria:

* Severe major depressive episode or significant autolytic ideation
* Showing symptoms of psychosis or substance abuse.
* If a participant relapses or progresses from her illness during the study period, the clinical psychologist responsible for the therapeutic group to which is assigned will ask the participant if they want to be referred to their hospital for individual psychological treatment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change in Posttraumatic Symptoms (patients) | Time 0 (baseline), Time 1 (change between Time 0 and post-intervention), Time 2 (change between T1 and 3 months post-intervention) and Time 3 (change between Time 2 and 12 months post-intervention)
  PCL-C (Posttraumatic Checklist -Civilian Version; Weathers et al., 1991), validated in Spanish for cancer patients (Costa-Requena and Gil, 2010). It assesses the presence of symptoms of posttraumatic stress.
Change in Posttraumatic Growth (patients) | Time 0 (baseline), Time 1 (change between Time 0 and post-intervention), Time 2 (change between T1 and 3 months post-intervention) and Time 3 (change between Time 2 and 12 months post-intervention)
  PTGI (Posttraumatic Growth Inventory; Tedeschi and Calhoun, 1996) validated in Spanish for patients with cancer (Costa-Requena and Gil, 2007).
Change in Distress (Anxiety and Depression) (patients) | Time 0 (baseline), Time 1 (change between Time 0 and post-intervention), Time 2 (change between T1 and 3 months post-intervention) and Time 3 (change between Time 2 and 12 months post-intervention)
  HADS (Hospital Anxiety and Depression Scale; Zigmond AS & Snaith, 1983), validated in Spanish for cancer patients (Costa-Requena et al., 2009). It assesses the levels of Anxiety and Depression in patients.
Change in Quality of Life (patients) | Time 0 (baseline), Time 1 (change between Time 0 and post-intervention), Time 2 (change between T1 and 3 months post-intervention) and Time 3 (change between Time 2 and 12 months post-intervention)
  EuroQol 5D (EQ-5D) European Quality of Life Scale. Spanish version. (Abadia et al., 1999).

SECONDARY OUTCOMES:
Change in Healthy Life Style (patients) | Time 0 (baseline), Time 1 (change between Time 0 and post-intervention), Time 2 (change between T1 and 3 months post-intervention) and Time 3 (change between Time 2 and 12 months post-intervention)
  Healthy lifestyles. It will be assessed through the Self-Report of Non-Healthy Habits. (Capdevila, 2005).
Perception of Social Support (patients) | Time 0 (baseline)
  MOS-SSS (Medical Outcomes Study Survey-Social Support; Sherbourne & Stewart, 1991) validated in Spanish for cancer patients (Costa, Salamero and Gil, 2007). It assesses the perception of social support.
Days of return-to-work (patients) | Time T1 (post-intervention) and Time 3 (12 months from T1)
  Work reincorporation. The following variables will be collected: number of days of sick leave until the return to work, changes of work and granting of total or absolute incapacity. It will be used the questionnaire devised by Nieuwenhuijsen et al. (2006) specifically to assess the return to work.
Fidelity to treatment (therapists) | Time 0 (baseline)
  Therapists´ fidelity to treatment will be assessed using the The Revised Cognitive Therapy Scale (CTS-R; Blackburn et al., 2000; James, Blackburn, & Reichelt, F, 2001)

OTHER OUTCOMES:
Time since diagnosis (patients) | Time 0 (baseline)
  Days since being diagnosed with breast cancer
Life Extreme Experiences (patients) | Time 0 (baseline)
  Inventory of Extreme Experiences (IEE) (Pérez-Sales, Cervellón, Vázquez, Vidales, and Gaborit, 2005): This instrument collects data from 34 experiences (most commonly related to trauma, loss or crisis, plus 5 vital positive events).
Biomarkers (patients) | Time 0 (baseline)
  For estrogen-alpha receptors (RE) a Dako monoclonal antibody Ref: IR657 / IS657. For progesterone receptors (RP) a Dako monoclonal antibody Ref: IR068 / IS068. For ki-67 a Dako monoclonal antibody Ref.IR626 / IS626. Finally, for Her-2 neu, herceptest Dako Ref.SK001.IR657/IS657. Para receptores de progesterona (RP) un anticuerpo monoclonal Dako Ref: IR068/IS068. Para ki-67 un anticuerpo monoclonal Dako Ref.IR626/IS626. Finalmente, para Her-2 neu, herceptest Dako Ref.SK001.

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Ochoa, PhD, Principal Investigator — Institut Català d'Oncologia
Locations (1):
- Institut Català d'Oncologia, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Ochoa C, Sumalla EC, Maté J, Castejón V, Rodríguez A, Blanco I, Gil F. Psicoterapia positiva grupal en cáncer. Hacia una atención psicosocial integral del superviviente de cáncer. Psicooncología 7(1):7-34, 2010.
- [Background] Ochoa C, Casellas-Grau A, Vives J, Font A, Borras JM. Positive psychotherapy for distressed cancer survivors: Posttraumatic growth facilitation reduces posttraumatic stress. Int J Clin Health Psychol. 2017 Jan-Apr;17(1):28-37. doi: 10.1016/j.ijchp.2016.09.002. Epub 2016 Oct 18. PMID 30487878
- [Derived] Lleras de Frutos M, Medina JC, Vives J, Casellas-Grau A, Marzo JL, Borras JM, Ochoa-Arnedo C. Video conference vs face-to-face group psychotherapy for distressed cancer survivors: A randomized controlled trial. Psychooncology. 2020 Dec;29(12):1995-2003. doi: 10.1002/pon.5457. Epub 2020 Aug 7. PMID 32618395